CLINICAL TRIAL: NCT03571178
Title: Quantitative Ultrasound of Trapezius Muscle in Cervical Myofascial Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09.2018.047
Record Dates: First submitted 2018-06-16; First posted 2018-06-27 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Myofascial Pain Syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Patients who will receive physical therapy
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — Physical therapy consisting of the application of hotpack, TENS and treatment ultrasound

SUMMARY:
The myofascial points within the trapezius muscle are hypoechogenic regions that can be depicted via ultrasound imaging. In this study we aimed to demonstrate the hypoechogenic regions within the trapezius muscle and to determine if physical therapy modalities change the appearance and size of these areas. We also wanted to explore if the presence of these areas correlate with pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with myofascial pain syndrome in the cervical region

Exclusion Criteria:

* Presence of cervical radiculopathies
* Previous history of cervical injusy
* Presence of rheumatologic diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | 3 weeks
  Pain

CONTACTS AND LOCATIONS:
Locations (1):
- Ozge Kenis Coskun, Istanbul, Kadikoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sancar M, Kenis-Coskun O, Gunduz OH, Kumbhare D. Quantitative Ultrasound Texture Feature Changes With Conservative Treatment of the Trapezius Muscle in Female Patients With Myofascial Pain Syndrome. Am J Phys Med Rehabil. 2021 Nov 1;100(11):1054-1061. doi: 10.1097/PHM.0000000000001697. PMID 33480607